CLINICAL TRIAL: NCT06525571
Title: Outcomes of High-risk Non-muscle Invasive Bladder Cancer Treated With Blue Light Resection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Photocure ASA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00442199
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: Blue light cystoscopy; Cysview
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester; Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Blue light Cystoscopy (Experimental): Patients with bladder tumors will undergo BLC TURBT
  Interventions: Drug: Cysview; Device: Karl Storz D-Light C Photodynamic Diagnostic (PDD) system
- White light Cystoscopy (Active Comparator): Patients with bladder tumors will undergo WLC TURBT
  Interventions: Device: Karl Storz D-Light C Photodynamic Diagnostic (PDD) system

INTERVENTIONS:
Drug: Cysview — Blue light cystoscopy uses hexyl aminolevulinate (HAL, branded in the United States as Cysview), a prodrug which accumulates in the bladder tumors and improves the tumor's visualization.
  Other Names: Hexyl aminolevulinate (HAL)
  Arms: Blue light Cystoscopy
Device: Karl Storz D-Light C Photodynamic Diagnostic (PDD) system — Cystoscopy procedure
  Other Names: Cystoscopy equipment to detect Cysview uptake in the bladder tumors

SUMMARY:
Comparing white-light cystoscopy (WLC) and blue-light cystoscopy (BLC) in TURBT for high risk (HR) non-muscle invasive bladder cancer (NMIBC) patients is crucial to determine the most effective method for reducing residual disease burden and improving recurrence-free survival. Enhanced visualization with BLC may lead to more accurate resections, potentially decreasing recurrence rates and improving long-term outcomes for bladder cancer patients. Patients will be randomized to either WLC TURBT or BLC TURBT, and outcomes will be measured using standard-of-care testing with cystoscopy and cytology, along with minimal residual disease (MRD) burden evaluation using urine next-generation sequencing.

DETAILED DESCRIPTION:
Objectives are as follows:

Primary i) Comparison of the reduction in MRD burden score between pre-resection and post-resection urine samples across BLC and WLC resection arms of the study, and among patients with a high-grade tumor at time of resection ii) Comparison of the reduction in MRD burden score between pre-resection and post-resection urine samples across BLC and WLC resection arms of the study, and among all evaluable study participants.

Secondary i) Among all evaluable study participants: Recurrence-free survival (RFS) at 12 and 24 months using post-TURBT and three month surveillance urine sample time points in BLC and WLC arm.

ii) Among patients undergoing intravesical induction: Recurrence-free survival (RFS) at 12 and 24 months using post-TURBT and three month surveillance urine sample time points in BLC and WLC arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TURBT for radiographic or cystoscopic positive tumor
* 18+ years old
* Upper tract evaluated using standard of care throughout duration of the study
* Induction intravesical therapy initiated within four weeks of TURBT

Exclusion Criteria:

* Variant histology consisting of less than 50% urothelial carcinoma
* History, or current diagnosis, of upper tract tumor or muscle-invasive bladder cancer
* Prior history of pelvic radiation
* Active urinary tract infection (UTI)
* Patients who are noncompliant with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Residual disease burden | Up to 24 months
  The residual tumor burden will be assessed by the standard of care testing, such as cystoscopy and cytology at 3 month intervals.
Minimal residual disease burden | Up to 24 months
  Minimal residual disease (MRD) in urine will be measured utilizing the Convergent's UroAmp test at 3 month intervals.

SECONDARY OUTCOMES:
Recurrence-free survival | 24 months
  Recurrence-free survival rate will measured from the date of randomization to the first recurrence or to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Armine Smith, MD, Principal Investigator — Sibley Memorial Hospital
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No